CLINICAL TRIAL: NCT00004429
Title: Randomized Study of Recombinant Human Growth Hormone in Patients on Chronic Hemodialysis or Peritoneal Dialysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: FDA Office of Orphan Products Development (U.S. Federal Agency)
Collaborators: Vanderbilt University (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 199/13377; VUMC-FDR000943
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2007-10

CONDITIONS: Kidney Failure, Chronic
Keywords: end stage renal disease; rare disease; renal and genitourinary disorders
MeSH Terms: conditions — Kidney Failure, Chronic; Rare Diseases; Urogenital Diseases | interventions — Growth Hormone

INTERVENTIONS:
Drug: growth hormone

SUMMARY:
OBJECTIVES:

I. Assess the clinical safety and long term effects of recombinant human growth hormone on a defined range of nutritional indices in malnourished chronic hemodialysis and continuous ambulatory peritoneal dialysis patients.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is a randomized, double blind, placebo-controlled, cross-over study.

Prior to randomization each patient's protein and calorie intake is assessed and optimized as possible. Patients are randomized to receive either placebo or recombinant human growth hormone subcutaneously every other day for 6 months. At the end of this 6 month period, patients undergo a 4 week washout period. After the washout period, patients are crossed-over to the alternate regimen for an additional 6 months followed by another 4 week washout period.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

* On hemodialysis or peritoneal dialysis for more than 3 months
* Optimally dialyzed (urea reduction ratio greater than 65%)
* Suboptimal nutritional status identified by one of the following criteria: -Protein catabolic rate less than 0.85 g/kg/d calculated by three point urea kinetic modeling on at least 2 occasions over the past 6 months -Progressive unintentional weight loss of more than 2.5% of the initial or ideal body weight and/or patient weighs less than 90% of ideal body weight -Biochemical parameters of malnutrition defined by two or more of the following measurements over the past 3 months: Serum albumin no greater than 3.7 g/dL Serum transferrin concentration less than 250 mg/dL Serum prealbumin concentration less than 30 mg/dL Serum IGF-1 concentration less than 0.250 mg/mL

--Patient Characteristics--

* No active autoimmune, inflammatory, or infectious disease At least 6 months since any documented malignancy
* No unusual dietary restrictions At least 3 months since peritonitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 1999-12; Study Completion 2005-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Talat Alp Ikizler, Study Chair — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States